CLINICAL TRIAL: NCT00990678
Title: Study of Vitamin D Supplementation to Male HIV Sero-positive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Ulrich Bang, M.D., Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HH-JEBJ-HIVstudy; EudraCT 2006-005039-40; Danish Health 2612-3303
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: HIV Seropositive
Keywords: HIV-1; humans; vitamin D; 1-hydroxy-vitamin D; Rocaltrol; calcium; complementary therapies
MeSH Terms: conditions — HIV Seropositivity | interventions — Calcitriol; Vitamin D; Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- "Strong vitamin D" (Experimental): Calcium 400 Mg + Vitamin D3 10 microg, 3 times daily Rocaltrol 1.25 mg to 2.5 mg daily
  Interventions: Drug: Rocaltrol; Drug: Vitamin D; Drug: Calcium
- Vitamin D (Active Comparator): calcium 400 mg + 10 microgram Vitamin D3, 3 times daily
  Interventions: Drug: Vitamin D; Drug: Calcium
- Calcium (Placebo Comparator): Tablet Calcium 400 mg x 3 daily
  Interventions: Drug: Calcium

INTERVENTIONS:
Drug: Rocaltrol — tablet, Vitamin 1-OH-D3, total 1.25-2.5 mg daily
  Arms: "Strong vitamin D"
Drug: Vitamin D — tablets, vitamin D3, 30 microgram daily
  Arms: "Strong vitamin D"; Vitamin D
Drug: Calcium — tablets, 400 mg calcium, 3 times daily

SUMMARY:
The investigators want to investigate if HIV sero-positive males benefit from vitamin D supplementation. The study runs in 16 weeks and the participants are treated with one of three placebo controlled regimes (tablets):

1. Calcium
2. Calcium and 25-hydroxy-vitamin D
3. Calcium and 25-hydroxy-vitamin D and 1,25-dihydroxyvitamin D

The endpoints are:

* Serum vitamin D
* Parathyroid hormone
* ionized calcium
* T-lymphocyte fractions (naïve, mature, Tregs)
* Osteocalcin (bone metabolism)

ELIGIBILITY:
Inclusion Criteria:

* male
* HIV-positive
* at least 18 years old
* receiving HiglyActiveAntiRetroviral Therapy (HAART)

Exclusion Criteria:

* hypercalcemia
* tuberculosis
* osteoporosis or other bone disease
* cancer with bone metastasis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2010-02 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
serum-vitamin D metabolites | week 0
serum-vitamin D metabolites | week 2
serum-vitamin D metabolites | week 4
serum-vitamin D metabolites | week 8
serum-vitamin D metabolites | week 12
serum-vitamin D metabolites | week 16

SECONDARY OUTCOMES:
T-lymphocyte fractions Parathyroid hormone ionized calcium | week 0
T-lymphocyte fractions Parathyroid hormone ionized calcium | week 2
T-lymphocyte fractions Parathyroid hormone ionized calcium | week 4
T-lymphocyte fractions Parathyroid hormone ionized calcium | week 8
T-lymphocyte fractions Parathyroid hormone ionized calcium | week 12
T-lymphocyte fractions Parathyroid hormone ionized calcium | week 16

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich C Bang, M.D., Principal Investigator — Dept. of Endocrinology, Hvidovre Hospital
Locations (1):
- Dept. of endocrinology, Hvidovre Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Bang U, Kolte L, Hitz M, Dam Nielsen S, Schierbeck LL, Andersen O, Haugaard SB, Mathiesen L, Benfield T, Jensen JE. Correlation of increases in 1,25-dihydroxyvitamin D during vitamin D therapy with activation of CD4+ T lymphocytes in HIV-1-infected males. HIV Clin Trials. 2012 May-Jun;13(3):162-70. doi: 10.1310/hct1303-162. PMID 22592096